CLINICAL TRIAL: NCT03307044
Title: Fractional CO2 Laser Therapy for Survivors of Breast Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison Quick, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-17153; NCI-2017-01554 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-08-31; First posted 2017-10-11 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Breast Carcinoma; Cancer Survivor; Cervical Carcinoma; Dyspareunia; Vaginal Dryness
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Dyspareunia | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fractional CO2 laser therapy) (Experimental): Patients undergo fractional CO2 laser therapy every 4-6 weeks for 3 treatments.
  Interventions: Procedure: Laser Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Laser Therapy — Undergo fractional CO2 laser therapy
  Other Names: Therapy, Laser
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well fraction carbon dioxide (CO2) laser therapy works in treating vaginal atrophy in patients with breast cancer. Fraction CO2 laser therapy uses intense beams of light to cut, burn, or destroy tissue and may remodel vaginal tissue and direct controlled thermal damage of vaginal mucosa.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the feasibility of fractionated CO2 laser treatments in patients with breast cancer with vaginal atrophy by determining treatment completion rates and tolerability of treatment.

II. To demonstrate the efficacy of fractionated CO2 laser treatments in patients with breast cancer with vaginal atrophy as determined by improvement from baseline to post treatment in the score of the Vaginal Assessment Scale (VAS).

SECONDARY OBJECTIVES:

I. Sexual behavior/function as measured by the Sexual Experiences Scare, Global sexual satisfaction scale, Female Sexual Function Index (FSFI), and the Female Sexual Distress Scare (FSDS).

II. Other symptoms of urogenital atrophy using the Urogenital Distress Inventory (UDI).

III. Overall patient assessment of symptoms by Patient Global Impression of Improvement scale (PGI-I).

OUTLINE:

Patients undergo fractional CO2 laser therapy every 4-6 weeks for 3 treatments.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with non-metastatic breast cancer with any hormone receptor and Her 2 neu status who have completed surgery, chemotherapy, and radiation and are currently on endocrine therapy, single agent Herceptin, or observation
* Symptoms of urogenital atrophy including dyspareunia or vaginal dryness

Exclusion Criteria:

* Patients with metastatic breast cancer
* Vaginal stenosis which would not allow vaginal probe to be placed (based on physician exam)
* Active genital infection at the time of enrollment (if present initially, can be treated and then patient can be re-evaluated for eligibility)
* Pelvic organ prolapse greater than stage II
* Prior reconstructive pelvic surgery involving mesh
* Hormone replacement therapy, vaginal estrogen therapy, DHEA, or biosynthetics within 6 weeks prior to enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Assessment Scale score | Baseline up to 4 weeks
  Using Vaginal Assessment Scale (VAS)
Patient compliance rates | Up to 4 weeks
  Compliance rates with treatment will be assessed.
Feasibility of laser treatments defined by completion rates and tolerability of treatment | Up to 4 weeks
  Will evaluate if laser can be completed and tolerated will be used to summarize demographics and clinical characteristics.

SECONDARY OUTCOMES:
Other symptoms of urogenital atrophy using the Urogenital Distress Inventory | Up to 4 weeks
  Descriptive statistics will be used to summarize demographics and clinical characteristics. Will either compare categorical responses from baseline to post treatment using McNemars Chi-square test or compare the change in response using a Signed Rank Test. Data will be transformed or a nonparametric test will be conducted if necessary.
Sexual behavior/function as measured by the Sexual Experiences Scare, Global sexual satisfaction scale, Female Sexual Function Index, and the Female Sexual Distress Scare | Up to 4 weeks
  Descriptive statistics will be used to summarize demographics and clinical characteristics. Will either compare categorical responses from baseline to post treatment using McNemar?s Chi-square test or compare the change in response using a Signed Rank Test. Data will be transformed or a nonparametric test will be conducted if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Quick, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu